CLINICAL TRIAL: NCT03753672
Title: Central Venous Pressure (CVP) Changes do Not Predict Preload Unresponsiveness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital Antoine Beclere (Other)
Responsible Party: Principal Investigator, Hamzaoui Olfa, principal investigator, Hopital Antoine Beclere
Other Study IDs: 2017-A03578-45
Record Dates: First submitted 2018-11-19; First posted 2018-11-27 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Cardiovascular Shock
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preload responsive: defined as an increase in Velocity time integral of the sub-aortic flow greater or equal to 10%
  Interventions: Diagnostic Test: preload responsiveness
- preload unresponsive: defined as an increase in Velocity time integral of the sub-aortic flow lower than 10%
  Interventions: Diagnostic Test: preload responsiveness

INTERVENTIONS:
Diagnostic Test: preload responsiveness — We investigated whether an increase in CVP ≥ 5 mmHg during PLR predict preload unresponsiveness diagnosed by the absence of increase in velocity-time integral (VTI) of the flow in the left ventricular outflow tract by more than 10%

SUMMARY:
Passive leg raising (PLR) is routinely used to predict preload responsiveness in critically ill patients. However, real-time measurements of cardiac output are required to assess its effects. Some authors have suggested that in fluid non-responders, central venous pressure (CVP) increased markedly. By analogy with the CVP rules proposed by Weill et al to assess a fluid challenge, it has been hypothesized that an increase in CVP ≥ 5 mmHg during PLR can predict preload unresponsiveness.

Objective Investigation of whether an increase in CVP ≥ 5 mmHg during PLR predict preload unresponsiveness diagnosed by the absence of increase in velocity-time integral (VTI) of the flow in the left ventricular outflow tract by more than 10% (4).

Methods Critically ill patients with a central venous catheter in place and for whom the physician decided to test preload responsiveness by PLR were prospectively included. Transthoracic echocardiography was performed to obtain VTI. The CVP and VTI were measured before and during PLR.

ELIGIBILITY:
Inclusion Criteria:

* ADULTS
* Patients presenting with shock or other signs of circulatory failure (tachycardia, oliguria)
* Need for the physician to test preload responsiveness
* Patients already equipped by a central venous catheter for the measurement of CVP

Exclusion Criteria:

* patients<18 years old
* pregnancy
* instaility justifying rapid increase in cathecolamines

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients with a central venous catheter in place and for whom the physician decided to test preload responsiveness by PLR were prospectively included. Transthoracic echocardiography was performed to obtain VTI. The CVP and VTI were measured before and during PLR.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2017-12-10 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
the predictive value of changes in CVP to determine preload responsiveness | ONE MINUTE TEST
  Systolic, diastolic and mean arterial pressure will be assessed before and after the PLR test

CONTACTS AND LOCATIONS:
Locations (1):
- Hamzaoui Olfa, Clamart, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hamzaoui O, Gouezel C, Jozwiak M, Millereux M, Sztrymf B, Prat D, Jacobs F, Monnet X, Trouiller P, Teboul JL. Increase in Central Venous Pressure During Passive Leg Raising Cannot Detect Preload Unresponsiveness. Crit Care Med. 2020 Aug;48(8):e684-e689. doi: 10.1097/CCM.0000000000004414. PMID 32697509